CLINICAL TRIAL: NCT01326910
Title: A Double-Blind, Randomized, Active-Controlled Clinical Trial to Evaluate the Efficacy and Safety of an Over-the-Counter Cream in the Management of Mild to Moderate Atopic Dermatitis in Children
Brief Title: Human Testing of an Over-the-Counter (OTC) Cream in Children With Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Products Company Division of Johnson & Johnson Consumer Companies, Inc. (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COOADM3002; HTR 11-130435-111 (Other: CRO)
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-06

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 19306-127 (Experimental): Experimental Topical cream applied twice daily (or as needed)
  Interventions: Drug: Colloidal Oatmeal
- 19306-137 (Other): Marketed Topical cream applied twice daily (or as needed)
  Interventions: Device: Topical Cream

INTERVENTIONS:
Drug: Colloidal Oatmeal — Topical cream applied twice daily (or as needed)
  Other Names: Not yet marketed
  Arms: 19306-127
Device: Topical Cream — Topical cream applied twice daily (or as needed)
  Other Names: EpiCeram
  Arms: 19306-137

SUMMARY:
This three week study will be conducted to determine the safety and efficacy of an over-the-counter (OTC) cream in children with mild to moderate atopic dermatitis.

DETAILED DESCRIPTION:
The objective of this trial is to evaluate the efficacy and safety of an OTC colloidal oatmeal skin protectant cream in children with mild to moderate AD in comparison to that of EpiCeram®

ELIGIBILITY:
Inclusion Criteria:

* Children ages 6 mo- 18 years
* Any ethnicity
* Diagnosed with atopic dermatitis (AD) per Hanifin-Rajka criteria
* Mild to moderate atopic dermatitis per Rajka-Langeland severity index
* Willing to use only provided cream and body wash for duration of study

Exclusion Criteria:

* Known sensitivity to investigational products
* Pregnant or breastfeeding
* Severe AD per Rajka-Langeland severity index
* AD requiring class I (super potent) or class II or III (potent) topical steroids
* Requires greater than 2.0 g inhaled or intranasal corticosteroids
* Other skin conditions which may interfere with the scoring of AD

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2011-03; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Qing Li, MD, PhD, Study Director — Johnson & Johnson Consumer and Personal Products Worldwide
Locations (2):
- United States (2):
  - Hilltop Research, St. Petersburg, Florida
  - Hilltop Research, Miamiville, Ohio

REFERENCES:
- [Derived] Lisante TA, Nunez C, Zhang P. Efficacy and safety of an over-the-counter 1% colloidal oatmeal cream in the management of mild to moderate atopic dermatitis in children: a double-blind, randomized, active-controlled study. J Dermatolog Treat. 2017 Nov;28(7):659-667. doi: 10.1080/09546634.2017.1303569. Epub 2017 Apr 2. PMID 28366039

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 19306-127 | 19306-137
Started | 45 | 45
Completed | 41 | 42
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 19306-127 | 19306-137 | Total
Number analyzed (Participants) | 45 | 45 | 90
Age Continuous [Mean (Standard Deviation); unit: years] | 6.9 (3.26) | 9.3 (4.26) | 8.1 (3.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 22 | 19 | 41
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Eczema Area and Severity Index (EASI)
Description: A regional body surface area tabulation based on severity ranging from 0 (none) to 3 (severe), and severity of signs of disease, then multiplied by body area with final calculation ranging from 0-72
Time Frame: 3 weeks
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 19306-127 | 19306-137
Number analyzed (Participants) | 45 | 45
units on a scale
  Day 0, Baseline | 3.014 (1.9473) | 3.359 (3.6925)
  Day 7, Week 1 | 1.286 (1.0137) | 1.621 (1.9275)
  Day 14, Week 2 | 1.310 (2.0153) | 1.298 (1.5811)
  Day 21, Week 3 | 1.154 (1.1570) | 1.064 (1.1320)

2. Secondary Outcome: Interim Eczema Area and Severity Index (EASI)
Description: Number of subjects improved at Week 2 compared to Baseline in EASI. Improved is defined as post baseline EASI score smaller than baseline score.
Time Frame: Week 2
Population: Intention to Treat
Measure: Number; unit: participants
Arm/Group | 19306-127 | 19306-137
Number analyzed (Participants) | 41 | 42
participants
  Improved | 38 (1.8789) | 38 (2.8447)
  Not Improved | 3 | 4

3. Secondary Outcome: Assessment of Itch
Description: Subject's or caregiver's assessment of itch, on a 10-cm Visual Analogue Scale (VAS), where 0-no itch, 10-worst itch imaginable
Time Frame: through Week 3
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 19306-127 | 19306-137
Number analyzed (Participants) | 45 | 45
units on a scale
  Day 0, Baseline | 1.557 (2.2526) | 1.208 (2.4939)
  Day 7, Week 1 | 1.840 (2.2876) | 1.537 (2.2051)
  Day 14, Week 2 | 2.199 (2.4595) | 1.480 (2.1464)
  Day 21, Week 3 | 1.972 (2.7890) | 1.685 (2.5902)

4. Secondary Outcome: Investigator's Global Atopic Dermatitis Assessment (IGADA)
Description: An assessment of Atopic Dermatitis based on a 4 point scale where 0 (none) and 3 (severe) are used to describe signs and symptoms in 4 designated body regions. Based on the presence or absence of the total number of signs and symptoms, the final rating will be 0-clear, 1-almost clear, 2-mild, 3-moderate, 4-severe, or 5-very severe.
Time Frame: through Week 3
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 19306-127 | 19306-137
Number analyzed (Participants) | 45 | 45
units on a scale
  Day 0, Baseline | 2.159 (0.6078) | 2.182 (0.6567)
  Day 7, Week 1 | 1.690 (0.6803) | 1.667 (0.7861)
  Day 14, Week 2 | 1.585 (0.7062) | 1.548 (0.8025)
  Day 21, Week 3 | 1.585 (0.8055) | 1.381 (0.7949)

ADVERSE EVENTS:
Time Frame: Three Weeks plus 30 days for Serious Adverse Events
Arm/Group | 19306-127 | 19306-137
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 6/45 | 2/45
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 19306-127 (N=45) | 19306-137 (N=45)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 1
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 1 | 0
PYREXIA (General disorders) | 2 | 0
SEASONAL ALLERGY (Immune system disorders) | 1 | 0
EAR INFECTION (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The trial was conducted as work made for hire, and disclosure of results by the investigator is prohibited without the prior written consent of Sponsor.